### INFORMED CONSENT FORM

### PATIENTS AND NURSING STAFF

# The impact of gaming on functioning among people with schizophrenia: a randomised controlled trial (GAME-A)

NCT number: NCT05707689

Date of the document: 15 February 2023

#### SUBJECT'S CONSENT TO PARTICIPATE IN THE STUDY (PATIENT)

# The impact of gaming on functioning among people with schizophrenia: a randomised controlled trial (GAME-A)

I have been asked to participate in the above-mentioned scientific study, which aims to assess the effects of computer gaming on functioning, symptoms, self-resilience, quality of life, acceptability of intervention and possible adverse effects in people with psychotic disorders. I understand that the gaming intervention is intended for the research participants only. I am also aware that the computer gaming intervention will last for a total of 10 weeks. It will take place 2 times a week, for about 60 minutes at a time (20 hours in total). The games will be played on the premises of the research organisations. The computer game to be played is an entertaining, non-violent multiplayer game. The game will be played in small groups, with a maximum of 8 participants per group. Participants will have access to University of Turku laptops, on which the game will already be installed. I am aware that a game instructor will be present during the game sessions to supervise the gaming and to help with any problems that may arise during the game. There is no cost to the player for using the game.

I have read and understood the research information, and I give my informed consent to participate in the study. I have been adequately informed about the study and the collection, processing and disclosure of data to be carried out in connection with the study. I understand that, upon giving my consent, my name, telephone number and email address will be collected. I understand that I will be contacted (phone call/text message/email/letter) in connection with research and data collection.

I am aware that my background information (age, gender, marital status, highest level of education, employment status, housing status, number of psychiatric hospitalisations and age at first contact with the psychiatric health care system), the questionnaires I have completed, a questionnaire to assess my functional capacity (PSP) completed by the nursing staff, the adverse effects form completed by the gaming instructor, and my diary of my gaming experiences and the amount of gaming I have done will be used in the study. At baseline, providing the background information and completing the questionnaires will take about 20-28 minutes per participant. After three and six months from the time I give my consent, it will take approximately 20-26 minutes/participant/survey session to complete the questionnaires. I am aware that the nursing staff at the research centres of the City of Helsinki and Central Finland Hospital District will assess and complete the questionnaire to assess my functional capacity (PSP) at baseline and after three and six months from the date of giving my consent. This will take less than 5 minutes of nursing staff time per participant. In addition, I am aware that the game instructor will fill out an adverse effects form for any adverse events that I may experience during the intervention. The information on adverse effects may be based on information provided by the nursing staff, descriptions that I provide or the game instructor's own observations during the game sessions. I understand that the game instructor will collect information from me and/or the nursing staff about possible adverse effects (e.g., changes in medication dosage, psychological symptoms and changes, psychiatric hospitalisations,

different forms of violence and serious side effects). I am aware that the data will be collected and processed as part of the study between 14 December 2022 and 31 December 2024.

I am also aware that the nursing staff will assess my eligibility for the study on the basis of the following information from the personal data register or patient information system: diagnosis of psychotic disorder (F20 to F29, ICD-10), age, diagnosis of major depression, mania or hypomanic episode, or developmental disability (ICD-10), severe visual impairment, diagnosis of gaming addiction or signs of that, substance abuse (other than nicotine addiction), head injury, hemiplegia or other neurological disease, or receiving electroconvulsive therapy (ECT) in the past six months.

I also understand that the nursing staff will assess whether I am proficient in Finnish, able to make my own decisions about my participation in the study, and able to give my written informed consent (no appointed guardian). This information will be used to assess the inclusion and exclusion criteria of the study. I am also aware that my participation in the study may be refused if the nursing staff consider that my participation would cause me harm.

I have had the opportunity to receive additional information about the study orally, and I have received adequate answers to all my questions about the study.

I have had sufficient time to consider taking part in the study. I have been adequately informed about the purpose and conduct of the study, the benefits and risks of the study, and my rights. I have not been pressured or tempted to take part in the study. I am also aware that I have been confirmed by the organisation's nursing staff as meeting the inclusion criteria for the study.

I am aware that my data will be treated confidentially by the members of the research team and will not be disclosed to another register or to another processor. The research material will not be disclosed to any person outside of this research. Furthermore, my data will not be transferred outside the EU or EEA (European Economic Area).

I understand that the research material I produce will only be used for the purposes of this study. I am aware that my personal data may also be processed in the context of an inspection by a domestic or foreign authority, a regular quality control of the research by a person who is not part of the research team (research monitor) and/or a quality assurance activity carried out by a representative of the commissioner.

I am aware that the results of the research will be reported and published locally through national and regional seminars, social media, professional publications and news on the study subject. In addition, four scientific publications will be submitted to high quality journals, and oral presentations will be given at national and international conferences. One doctoral dissertation will also be conducted based on the research.

I understand that participation in this study is voluntary. I understand that I have the right to refuse to participate in the study. I may also discontinue my participation in the study or

withdraw my consent later at any stage of the study without giving any reason. If I wish to withdraw my participation in the study, I can inform the researcher at the Department of Nursing at the University of Turku (050-4766116, <a href="maijakatriina.satamo@utu.fi">maijakatriina.satamo@utu.fi</a>) of my decision. I am aware that if I discontinue participation in the study or withdraw my consent and participation in the study, the data collected about me up to the point of discontinuation and withdrawal of consent will be used as part of the study. After the study concludes, the data containing my personal information will be stored for 15 years, after which it will be destroyed. I understand that I will not be reimbursed for any expenses incurred for participating in the study. Refusing to participate in the study or withdrawal of consent will not have negative consequences or affect my treatment, care or access to services.

| I confirm my participation in this study, and I voluntarily agree to be a research subject. |
|---|
| Signature: |
| Printed name and date: |
| E-mail address and telephone number: |
| Contact details of the person(s) receiving the consent: |
| Researcher Christa Erkkilä, <u>christa.erkkila@utu.fi</u> |
| Researcher Maija Satamo, maijakatriina.satamo@utu.fi, tel. 050 476 6116 |
| The person in charge of the study, Professor Maritta Välimäki, <u>mava@utu.fi</u> (in special circumstances where researchers are unable to collect patient consent within the organisation). |
| Signature and name clarification of the person receiving the consent, and date: |

A copy of the document will be given to the person giving consent.

## TUTKITTAVAN SUOSTUMUS TUTKIMUKSEEN OSALLISTUMISESTA (ASIAKAS)

## Tietokonepelien vaikutus skitsofreniaa sairastavan potilaan toimintakykyyn: satunnaistettu kontrolloitu tutkimus (GAME-A)

Minua on pyydetty osallistumaan yllä mainittuun tieteelliseen tutkimukseen, jonka tarkoituksena on selvittää pelaamisen vaikutuksia psykoottista häiriötä sairastavien henkilöiden toimintakykyyn, oireisiin, minäpystyvyyteen, elämänlaatuun, intervention hyväksyttävyyteen sekä mahdollisiin haittavaikutuksiin. Ymmärrän, että peli-interventio on tarkoitettu vain tutkimukseen osallistujille. Tiedostan myös, että tietokonepeli-interventio kestää yhteensä 10 viikkoa. Se toteutetaan 2 kertaa viikossa, noin 60 minuuttia kerrallaan (yhteensä 20 tuntia). Pelaaminen toteutetaan tutkimusorganisaatioiden tiloissa. Pelattava tietokonepeli on viihdyttävä moninpeli, joka ei sisällä väkivaltaa. Pelaaminen toteutetaan pienryhmissä, maksimissaan 8 osallistujaa per ryhmä. Osallistujilla on käytössään Turun yliopiston kannettavat tietokoneet, joihin peli on asennettu valmiiksi. Tiedän, että pelihetkiin osallistuu peliohjaaja, joka valvoo pelaamisen toteutumista ja auttaa mahdollisissa pelaamiseen liittyvissä ongelmatilanteissa. Pelien käytöstä ei aiheudu pelaajalle kustannuksia.

Olen lukenut ja ymmärtänyt saamani tutkimustiedotteen ja annan tietoon perustuvan suostumukseni tutkimukseen. Olen saanut riittävästi tietoa tutkimuksesta ja sen yhteydessä suoritettavasta tietojen keräämisestä, käsittelystä ja luovuttamisesta. Ymmärrän, että suostumusta annettaessa minulta kerätään nimi, puhelinnumero sekä sähköpostiosoite. Ymmärrän, että minuun ollaan yhteydessä (puhelu/tekstiviesti/sähköposti/kirje) tutkimukseen ja aineistonkeruuseen liittyen.

Olen tietoinen, että taustatietojani (ikä, sukupuoli, siviilisääty, korkein koulutustaso, työllisyystilanne, asumistilanne, psykiatristen sairaalahoitojaksojen määrä sekä ikä kontaktissa ensimmäisessä psykiatrisen terveyden-huoltojärjestelmän tuottamaani kyselyaineistoa, hoitohenkilökunnan täyttämää toimintakykyäni arvioivaa kyselyaineistoa (PSP), peliohjaajan täyttämää haittavaikutuslomaketta sekä päiväkirjaani pelikokemuksistani ja pelaamisen määrästä käytetään tutkimuksessa. Alkukartoituksessa taustatietoihin ja kyselylomakkeisiin vastaaminen vie aikaa noin 20–28 minuuttia/osallistuja. Kolmen ja kuuden kuukauden jälkeen potilaan suostumuksen antamisesta kyselylomakkeisiin vastaaminen vie aikaa noin 20–26 minuuttia/osallistuja/kyselykerta. Olen tietoinen, että hoitohenkilökunta Helsingin ja Keski-Suomen sairaanhoitopiirin tutkimuskeskuksissa arvioi ja täyttää toimintakykyäni arvioivan kyselyn (PSP) alkukartoituksessa sekä kolmen ja kuuden kuukauden jälkeen potilaan suostumuksen antamisesta. Tämä vie hoitohenkilökunnan aikaa alle 5 minuuttia per osallistuja. Lisäksi olen tietoinen, että peliohjaaja täyttää haittavaikutuslomakkeen osallistujan mahdollisista intervention aikana haittavaikutuksista. Tiedot haittavaikutuksista voivat perustua hoitohenkilökunnan antamiin tietoihin, potilaan tuottamiin kuvauksiin tai peliohjaajan omiin havaintoihin pelikertojen aikana. Ymmärrän, että peliohjaaja kerää mahdollisista haittavaikutuksista tietoa minulta ja/tai hoitohenkilökunnalta (esim. lääkeannoksen muutokset, psyykkiset oireet ja niissä tapahtuvat

muutokset, psykiatriset sairaalajaksot, eri väkivallan muodot ja vakavat haittavaikutukset). Olen tietoinen, että tutkimuksessa tietoja kerätään ja käsitellään aikavälillä 14.12.2022 - 31.12.2024.

Lisäksi olen tietoinen, että hoitohenkilökunta arvioi sopivuuteni tutkimukseen henkilötietorekisteristä tai potilastietojärjestelmästä seuraavien tietojen perusteella: diagnoosi psykoottisesta häiriöstä (F20–F29, ICD-10), ikä, diagnoosi vakavasta masennuksesta, manialle tai hypomaaniselle jaksolle tai kehitysvammaisuuteen (ICD-10), vakava näkövamma, diagnoosi peliriippuvuudesta tai merkkejä siitä, päihteiden väärinkäyttö (muu kuin nikotiiniriippuvuus), päävamma, toispuolihalvaus tai muu neurologinen sairaus tai sähköhoidon saaminen (ECT) viimeisen kuuden kuukauden aikana.

Ymmärrän myös, että hoitohenkilökunta arvioi, olenko suomen kielen taitoinen, kykeneväinen päättämään omasta osallistumisestani tutkimukseen sekä antamaan kirjallisen tietoon perustuvan suostumukseni (ei määrättyä edunvalvojaa). Näitä tietoja käytetään tutkimuksen sisäänotto- ja poissulkukriteerien arvioimiseksi. Lisäksi tiedostan, että tutkimukseen osallistumiseni voidaan evätä, jos hoitohenkilökunta arvioi osallistumisen aiheuttavan minulle haittaa.

Minulla on ollut mahdollisuus saada suullisesti lisätietoa tutkimuksesta ja olen saanut riittävän vastauksen kaikkiin tutkimusta koskeviin kysymyksiini.

Minulla on ollut riittävästi aikaa harkita tutkimukseen osallistumista. Olen saanut riittävät tiedot tutkimuksen tarkoituksesta ja sen toteutuksesta, tutkimuksen hyödyistä ja riskeistä sekä oikeuksistani. Minua ei ole painostettu eikä houkuteltu osallistumaan tutkimukseen. Olen myös tietoinen siitä, että organisaation hoitohenkilökunta on vahvistanut minun täyttävän tutkimuksen sisäänottokriteerit.

Tiedän, että tutkimusryhmän jäsenet käsittelevät tietojani luottamuksellisesti eikä niitä luovuteta toiseen rekisteriin tai toiselle henkilötietojen käsittelijälle. Tutkimusaineistoa ei luovuteta tutkimuksen ulkopuolisille henkilöille. Tietojani ei myöskään siirretä EU:n tai ETAN ulkopuolelle.

Ymmärrän, että tuottamaani tutkimusmateriaalia käytetään ainoastaan tässä tutkimuksessa. Olen tietoinen siitä, että henkilötietojani voidaan käsitellä myös kotimaisen ja ulkomaisen viranomaisen suorittaman tarkastuksen, tutkimustiimiin kuulumattoman tutkimuksen säännönmukaista laadunvalvontaa tekevän henkilön ja/tai toimeksiantajan edustajan suorittaman laadunvarmistustoiminnan yhteydessä.

Olen tietoinen, että tutkimustulokset raportoidaan ja julkistetaan paikallisesti kansallisissa ja alueellisissa seminaareissa, sosiaalisessa mediassa sekä kirjoittamalla ammattijulkaisuja sekä uutisia aiheesta. Lisäksi neljä tieteellistä julkaisua toimitetaan korkealaatuisiin lehtiin sekä suullisia esityksiä pidetään kansallisissa ja kansainvälisissä konferensseissa. Tutkimuksen pohjalta laaditaan myös yksi väitöskirja.

Ymmärrän, että tähän tutkimukseen osallistuminen on vapaaehtoista. Olen selvillä siitä, että minulla on oikeus kieltäytyä tutkimukseen osallistumisesta. Voin myöhemmin halutessani myös keskeyttää osallistumiseni tutkimukseen tai peruuttaa antamani suostumus missä tahansa tutkimuksen vaiheessa syytä ilmoittamatta. Jos haluan peruuttaa tutkimukseen osallistumiseni, voin ilmoittaa päätöksestäni Turun yliopiston hoitotieteen laitoksen tutkijalle (050-4766116, maijakatriina.satamo@utu.fi). Olen tietoinen siitä, että mikäli keskeytän tutkimuksen tai peruutan suostumuksen, minusta keskeyttämiseen ja suostumuksen peruuttamiseen mennessä kerättyjä tietoja käytetään osana tutkimusta. Tutkimuksen päätyttyä henkilötietojani sisältävä aineisto säilytetään 15 vuotta, jonka jälkeen se tuhotaan. Tiedän, että tutkimukseen osallistumisesta aiheutuneista kuluista ei makseta korvausta. Tutkimuksesta kieltäytyminen tai suostumuksen peruuttaminen ei aiheuta kielteisiä seurauksia eikä se vaikuta kohteluuni, hoitooni tai palvelujen saantiini.

| Vahvistan osallistumiseni tähän tutkimukseen ja suostun vapaaehtoisesti tutkimushenkilöksi. |
|---|
| Allekirjoitus: |
| Nimenselvennys ja päivämäärä: |
| Sähköpostiosoite ja puhelinnumero: |
| Suostumuksen vastaanottavien henkilöiden yhteystiedot: |
| Tutkija Christa Erkkilä, <u>christa.erkkila@utu.fi</u> |
| Tutkija Maija Satamo, maijakatriina.satamo@utu.fi, p. 050 476 6116 |
| Tutkimuksesta vastaava henkilö, professori Maritta Välimäki, <u>mava@utu.fi</u> (erityisessä tilanteessa, mikäli tutkijat ovat estyneitä keräämään potilaiden suostumukset organisaatiossa) |
| Suostumuksen vastaanottavan henkilön allekirjoitus, nimenselvennys ja päivämäärä: |
| Jäljennös asiakirjasta annetaan suostumuksen antajalle. |

#### NURSING STAFF'S CONSENT TO PARTICIPATE IN THE STUDY

The impact of gaming on functioning among people with schizophrenia: a randomised controlled trial (GAME-A)

I have been asked to participate in the above-mentioned scientific study, which aims to assess the feasibility, acceptability and appropriateness of the intervention of gaming through interviews and questionnaires.

I have read and I understand the research information, and I give my informed consent to participate in the study. I have been adequately informed about the study and the collection, processing and disclosure of data to be carried out in connection with the study. I understand that, upon giving my consent, my name, telephone number and email address will be collected. I understand that I will be contacted (phone call/text message/email/letter) in connection with research and data collection. I am aware that my background information (age, gender, education, professional title, work experience in the social and health care sector) and the interview and survey data I provide will be used in the study. Providing the background information and completing the questionnaires and interview will take approximately 30–66 minutes per participant. I also understand that the interview will be recorded to increase the reliability of the analysis. I am aware that the data will be collected and processed as part of the study between 14 December 2022 and 31 December 2024.

I have had the opportunity to receive additional information about the study orally, and I have received adequate answers to all my questions about the study.

I have had sufficient time to consider taking part in the study. I have been adequately informed about the purpose and conduct of the study, the benefits and risks of the study, and my rights. I have not been pressured or tempted to take part in the study. I understand that any written, be it in electronic or paper form, and oral research material that I produce will be used only for the purpose of this study.

I am aware that my data will be treated confidentially by the members of the research team, and it will not be disclosed to another register or to another processor. The research material will not be disclosed to any person outside of this research. Furthermore, my data will not be transferred outside the EU or EEA (European Economic Area).

I understand that the research material I produce will only be used for the purposes of this study. I am aware that my personal data may also be processed in the context of an inspection by a domestic or foreign authority, a regular quality control of the research by a person who is not part of the research team (research monitor) and/or a quality assurance activity carried out by a representative of the commissioner.

I am aware that the results of the research will be reported and published locally through national and regional seminars, social media, professional publications and news on the study subject. In addition, four scientific publications will be submitted to high quality journals, and oral presentations will be given at national and international conferences. One doctoral dissertation will also be conducted based on the research.

I understand that participation in this study is voluntary. I understand that I have the right to refuse to participate in the study. I may also discontinue my participation in the study or withdraw my consent later at any stage of the study without giving any reason. If I wish to withdraw my participation in the study, I can inform the researcher at the Department of Nursing at the University of Turku (050-4766116, <a href="maijakatriina.satamo@utu.fi">maijakatriina.satamo@utu.fi</a>) of my decision. I am aware that if I discontinue participation in the study or withdraw my consent and participation in the study, the data collected about me up to the point of discontinuation and withdrawal of consent will be used as part of the study. After the study concludes, the data containing my personal information will be stored for 15 years, after which it will be destroyed. I understand that I will not be reimbursed for any expenses incurred for participating in the study. Refusing to participate in the study or withdrawal of consent will not have negative consequences or affect my treatment or position in the organisation.

| Pı | rinted name and date: |
|---|---|
| E | -mail address and telephone number: |
| C | ontact details of the person(s) receiving the consent: |
| R | esearcher Christa Erkkilä, <u>christa.erkkila@utu.fi</u> |
| R | esearcher Maija Satamo, maijakatriina.satamo@utu.fi, tel. 050 476 6116 |
| | he person in charge of the study, Professor Maritta Välimäki, <u>mava@utu.fi</u> (in sprcumstances where researchers are unable to collect patient consent within the organisat |
| Si | ignature and name clarification of the person receiving the consent, and date: |

I confirm my participation in this study, and I voluntarily agree to be a research subject.

#### HOITOHENKILÖKUNNAN SUOSTUMUS TUTKIMUKSEEN OSALLISTUMISESTA

### Tietokonepelien vaikutus skitsofreniaa sairastavan potilaan toimintakykyyn: satunnaistettu kontrolloitu tutkimus (GAME-A)

Minua on pyydetty osallistumaan yllä mainittuun tieteelliseen tutkimukseen, jossa arvioidaan intervention eli pelaamisen toteutettavuutta, hyväksyttävyyttä sekä sopivuutta haastattelun ja kyselyn avulla.

Olen lukenut ja ymmärtänyt saamani tutkimustiedotteen ja annan tietoon perustuvan suostumukseni tutkimukseen. Olen saanut riittävästi tietoa tutkimuksesta ja sen yhteydessä suoritettavasta tietojen keräämisestä, käsittelystä ja luovuttamisesta. Ymmärrän, että suostumusta annettaessa minulta kerätään nimi, puhelinnumero sekä sähköpostiosoite. Ymmärrän, että minuun ollaan yhteydessä (puhelu/tekstiviesti/sähköposti/kirje) tutkimukseen ja aineistonkeruuseen liittyen. Olen tietoinen, että taustatietojani (ikä, sukupuoli, koulutus, ammattinimike, työkokemus sosiaali- ja terveysalalla) sekä tuottamaani haastatteluja kyselyaineistoa käytetään tutkimuksessa. Taustatietoihin, kyselylomakkeisiin ja haastatteluun vastaaminen vie yhteensä aikaa noin 30-66 minuuttia per osallistuja. Lisäksi ymmärrän, että haastattelu nauhoitetaan analyysin luotettavuuden lisäämiseksi. Olen tietoinen, että tutkimuksessa tietoja kerätään ja käsitellään aikavälillä 14.12.2022 - 31.12.2024.

Minulla on ollut mahdollisuus saada suullisesti lisätietoa tutkimuksesta ja olen saanut riittävän vastauksen kaikkiin tutkimusta koskeviin kysymyksiini.

Minula on ollut riittävästi aikaa harkita tutkimukseen osallistumista. Olen saanut riittävät tiedot tutkimuksen tarkoituksesta ja sen toteutuksesta, tutkimuksen hyödyistä ja riskeistä sekä oikeuksistani. Minua ei ole painostettu eikä houkuteltu osallistumaan tutkimukseen. Ymmärrän, että tuottamaani kirjallista sähköisessä tai paperisessa muodossa sekä suullista tutkimusmateriaalia käytetään ainoastaan tässä tutkimuksessa.

Tiedän, että tutkimusryhmän jäsenet käsittelevät tietojani luottamuksellisesti eikä niitä luovuteta toiseen rekisteriin tai toiselle henkilötietojen käsittelijälle. Tutkimusaineistoa ei luovuteta tutkimuksen ulkopuolisille henkilöille. Tietojani ei myöskään siirretä EU:n tai ETAN ulkopuolelle.

Ymmärrän, että tuottamaani tutkimusmateriaalia käytetään ainoastaan tässä tutkimuksessa. Olen tietoinen siitä, että henkilötietojani voidaan käsitellä myös kotimaisen ja ulkomaisen viranomaisen suorittaman tarkastuksen. tutkimustiimiin kuulumattoman tutkimuksen säännönmukaista laadunvalvontaa tekevän henkilön toimeksiantajan edustajan ja/tai suorittaman laadunvarmistustoiminnan yhteydessä.

Olen tietoinen, että tutkimustulokset raportoidaan ja julkistetaan paikallisesti kansallisissa ja alueellisissa seminaareissa, sosiaalisessa mediassa sekä kirjoittamalla ammattijulkaisuja sekä uutisia aiheesta. Lisäksi neljä tieteellistä julkaisua toimitetaan korkealaatuisiin lehtiin sekä suullisia esityksiä pidetään kansallisissa ja kansainvälisissä konferensseissa. Tutkimuksen pohjalta laaditaan myös yksi väitöskirja.

Ymmärrän, että tähän tutkimukseen osallistuminen on vapaaehtoista. Olen selvillä siitä, että minulla on oikeus kieltäytyä tutkimukseen osallistumisesta. Voin myöhemmin halutessani myös keskeyttää osallistumiseni tutkimukseen tai peruuttaa antamani suostumus missä tahansa tutkimuksen vaiheessa syytä ilmoittamatta. Jos haluan peruuttaa tutkimukseen osallistumiseni, voin ilmoittaa päätöksestäni Turun yliopiston hoitotieteen laitoksen tutkijalle (050-4766116, maijakatriina.satamo@utu.fi). Olen tietoinen siitä, että mikäli keskeytän tutkimuksen tai peruutan suostumuksen ja osallistumiseni tutkimukseen, minusta keskeyttämiseen ja suostumuksen peruuttamiseen mennessä kerättyjä tietoja käytetään osana tutkimusta. Tutkimuksen päätyttyä henkilötietojani sisältävä aineisto säilytetään 15 vuotta, jonka jälkeen se tuhotaan. Tiedän, että tutkimukseen osallistumisesta aiheutuneista kuluista ei makseta korvausta. Tutkimuksesta kieltäytyminen tai suostumuksen peruuttaminen ei aiheuta kielteisiä seurauksia eikä se vaikuta kohteluuni tai asemaani organisaatiossa.

Vahvistan osallistumiseni tähän tutkimukseen ja suostun vapaaehtoisesti tutkimushenkilöksi.

Allekirjoitus:

Nimenselvennys ja päivämäärä:

Sähköpostiosoite ja puhelinnumero:

Suostumuksen vastaanottavien henkilöiden yhteystiedot:

Tutkija Christa Erkkilä, christa.erkkila@utu.fi

Tutkija Maija Satamo, maijakatriina.satamo@utu.fi, p. 050 476 6116

Tutkimuksesta vastaava henkilö, professori Maritta Välimäki, mava@utu.fi (erityisessä tilanteessa, mikäli tutkijat ovat estyneitä keräämään potilaiden suostumukset organisaatiossa)

Suostumuksen vastaanottavan henkilön allekirjoitus, nimenselvennys ja päivämäärä:

Jäljennös asiakirjasta annetaan suostumuksen antajalle.